CLINICAL TRIAL: NCT04693520
Title: A Phase 2, Single-arm Study of the Biomarker Effects of ALZ-801 in Subjects With Early Alzheimer's Disease Who Are Carriers of the ε4 Variant of the Apolipoprotein E Gene (APOE4/4 or APOE3/4)
Brief Title: Biomarker Effects of ALZ-801 in APOE4 Carriers With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alzheon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALZ-801-201ADBM
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Early Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ALZ-801

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental): ALZ-801 265 mg tablets once daily for two weeks and twice daily thereafter
  Interventions: Drug: ALZ-801

INTERVENTIONS:
Drug: ALZ-801 — ALZ-801 265 mg twice daily (BID)

SUMMARY:
The study will investigate the effects of oral ALZ-801, in subjects with Early AD who have the APOE4/4 or APOE3/4 genotype, on the biomarkers of core AD pathology. The objectives of this study include determining the efficacy and safety/tolerability of ALZ-801. In addition, the study will evaluate the extended PK profile over 8 hours in 16 subjects after 65 weeks of treatment.

DETAILED DESCRIPTION:
The LTE year 1 & 2 study will investigate the effects of oral ALZ-801, in subjects with Early AD who have the APOE4/4 or APOE3/4 genotype, on the biomarkers of core AD pathology. The objectives of LTE study are to continue longitudinal assessment of the efficacy and safety/tolerability of ALZ-801 over a total period of 4 years (2-year Core study plus 2 years of LTE).

Core study: ALZ-801 265 mg twice daily (BID) in the Core Study, Weeks 0-104

LTE year 1: ALZ-801 265 mg BID in the Core Study and the Long-Term Extension (LTE, Weeks 104-208)

LTE year 2: ALZ-801 265mg BID in the Core Study and LTE Year 1 (Weeks 104-156), and LTE Year 2 (Weeks 156-208)

ELIGIBILITY:
Inclusion Criteria

1. Age between 50 and 80 years, inclusive.
2. Early Alzheimer's Disease (AD): a diagnosis of Probable AD Dementia or Mild Cognitive Impairment (MCI) due to AD in accordance with the National Institute on Aging-Alzheimer's Association (NIA-AA) Working Group Criteria [Albert et al, 2011; McKhann et al, 2011].
3. One of the following apolipoprotein E (APOE) genotypes - either APOE4/4 (homozygous) or APOE3/4 (heterozygous).
4. MMSE score 22 to 30 inclusive; Clinical Dementia Rating (CDR)-Global Score of 0.5 or 1.0, and CDR Memory Box Score of ≥ 0.5.
5. Documented confirmation of AD diagnosis by either positive amyloid positron emission tomography (PET) or positive CSF AD signature. Subjects without documented positive AD biomarker status must have a positive CSF biomarker result from a sample provided at screening.
6. Stable doses of acetylcholinesterase for the duration of the study are allowed.

Exclusion Criteria

1. Brain MRI at screening indicative of significant abnormality
2. Diagnosis of neurodegenerative disorder other than AD
3. Current diagnosis of Major Depressive Disorder (MDD)
4. Concomitant treatment with memantine.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Plasma Biomarker of Core AD Pathology | Week 104
  Percent change from baseline in p-tau181
Incidence, Nature, and Severity of Treatment Emergent Adverse events (TEAE) | Week 108
  Safety and tolerability as measured by incidence, nature and severity of treatment emergent adverse events (TEAE), serious TEAE, and TEAE leading to withdrawal.
Volumetric Magnetic Resonance Imaging (vMRI) Biomarker - Hippocampal Volume | Weeks 104
  Change from baseline in hippocampal volume measured in mm3

SECONDARY OUTCOMES:
Plasma Biomarkers of AD and Neurodegeneration | Weeks 104
  Percent changes from baseline in: Aβ-40, Aβ-42,p-tau217 and plasma glial fibrillary acidic protein (GFAP),NfL
vMRI Biomarker - Ventricular volume and Cortical Thickness | Weeks 104, 156 and 208
  Change from baseline in cortical thickness measured in mm3
Additional CSF Biomarkers of AD Pathology and Neurodegeneration | Weeks 104
  Percent changes from baseline for: p-tau217,Aβ-40, Aβ-42, NfL, t-tau, sTREM2, YKL-40 and neurogranin
Incidence, Nature, and Severity of Treatment Emergent Adverse events (TEAE) | Week 160 and week 212
  Safety and tolerability as measured by incidence, nature and severity of treatment emergent adverse events (TEAE), serious TEAE, and TEAE leading to withdrawal.
Volumetric Magnetic Resonance Imaging (vMRI) Biomarker - Hippocampal Volume | Week 156 and week 208
  Change from baseline in hippocampal volume measured in mm3

OTHER OUTCOMES:
Cognitive assessment - Rey Auditory Verbal Learning Test (RAVLT) | Weeks 104, week 156 and week 208
  Change from baseline in RAVLT score
Cognitive Assessment - Digit Symbol Substitution Test (DSST) | Weeks 104, Week 156 and Week 208
  Change from baseline in DSST score
Functional Assessment - Amsterdam Instrumental Activities of Daily Living (A-IADL) | Weeks 104, Week 156 and Week 208
  Change from baseline in A-IADL score
Cognitive Assessment - Mini Mental State Examination (MMSE) | Weeks 104, Week 156 and Week 208
  Change from baseline in MMSE score
Global Assessment - Clinical Dementia Rating - Sum of Boxes (CDR-SB) | Weeks 104, Week 156 and Week 208
  Change from baseline in CDR-SB score

CONTACTS AND LOCATIONS:
Overall Officials: John Hey, PhD, Study Director — Alzheon Inc.
Locations (6):
- Czechia (3):
  - St. Anne's University Hospital, Brno
  - Motol University Hospital, Prague
  - Vestra Clinics, Rychnov nad Kněžnou
- Netherlands (3):
  - Brain Research Center, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - Brain Research Center, Zwolle

REFERENCES:
- [Derived] Hey JA, Yu JY, Abushakra S, Schaefer JF, Power A, Kesslak P, Paul J, Tolar M. Clinical Pharmacokinetics of Oral ALZ-801/Valiltramiprosate in a 2-Year Phase 2 Trial of APOE4 Carriers with Early Alzheimer's Disease. Clin Pharmacokinet. 2025 Mar;64(3):407-424. doi: 10.1007/s40262-025-01482-8. Epub 2025 Feb 5. PMID 39907966
- [Derived] Hey JA, Yu JY, Abushakra S, Schaefer JF, Power A, Kesslak P, Tolar M. Analysis of Cerebrospinal Fluid, Plasma beta-Amyloid Biomarkers, and Cognition from a 2-Year Phase 2 Trial Evaluating Oral ALZ-801/Valiltramiprosate in APOE4 Carriers with Early Alzheimer's Disease Using Quantitative Systems Pharmacology Model. Drugs. 2024 Jul;84(7):825-839. doi: 10.1007/s40265-024-02068-7. Epub 2024 Jun 20. PMID 38902572
- [Derived] Hey JA, Abushakra S, Blennow K, Reiman EM, Hort J, Prins ND, Sheardova K, Kesslak P, Shen L, Zhu X, Albayrak A, Paul J, Schaefer JF, Power A, Tolar M. Effects of Oral ALZ-801/Valiltramiprosate on Plasma Biomarkers, Brain Hippocampal Volume, and Cognition: Results of 2-Year Single-Arm, Open-Label, Phase 2 Trial in APOE4 Carriers with Early Alzheimer's Disease. Drugs. 2024 Jul;84(7):811-823. doi: 10.1007/s40265-024-02067-8. Epub 2024 Jun 20. PMID 38902571